CLINICAL TRIAL: NCT06143085
Title: Impact of Nonsurgical Periodontal Therapy for Stage 2 and 3 Periodontitis on Oral Health Related Quality of Life: A Clinical Trial
Brief Title: Impact of Nonsurgical Periodontal Therapy on Oral Health Related Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ali A Abdulkareem, Assistant Professor, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 663622
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Generalized periodontitis (Experimental): Patients diagnosed with generalized periodontitis of different severities exhibiting periodontal pockets not exceeding 6mm.
  Interventions: Procedure: Root surface debridement

INTERVENTIONS:
Procedure: Root surface debridement — Periodontitis patients are treated non-surgically by supra- and subgingival debridement followed by root surface debridement for moderately deep periodontal pockets (4 to 6mm)

SUMMARY:
Periodontitis is a destructive inflammatory disease of tooth supporting tissues and it adversely affects oral and general health as well as lowering the quality of life. Nonsurgical periodontal therapy is a gold standard technique for treating mild to moderate periodontitis and it was reported to significantly improve oral health related quality of life.

DETAILED DESCRIPTION:
Periodontitis is a chronic disease characterized by progressive loss of tooth-supporting tissues. It is adversely affecting function, esthetic, and general wellbeing. Oral health related quality of life (OHRQoL) is the part of quality of life which is affected by oral cavity-related status. Majority of clinical studies emphasize on periodontal outcomes after periodontal therapy. However, tangible outcomes perceived by the patient such as need for re-treatment, tooth survival, and OHRQoL are mostly neglected. OHRQoL is mainly measured by using self-reported questionnaires and the most commonly used one is Oral Health Impact Profile (OHIP).

Nonsurgical periodontal therapy (NSPT) is the gold-standard technique for treating shallow to moderately deep periodontal pockets. The principle of this technique is based on mechanically disrupting subgingival dysbiotic biofilm, consequently; restoring homeostasis and healthy state of periodontal tissues. Indeed, halting progressive periodontitis is a major contributor for improving oral health and increasing tooth survival rate which are positively perceived by the patients. Previous studies consistently reporting improvement of OHRQoL following periodontal treatment. Therefore, this study aimed to investigate the impact of NSPT on OHRQoL for Stage (S)2 and S3 periodontitis patient and the factors predicting the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Not reporting history of any systemic disease
* Non-smoker
* Can read and understand the questionnaire.

Exclusion Criteria:

* Patients with depression or any psychological issues
* Those not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth | PPD is assessed at baseline and 3 months after treatment
  The distance from the gingival margin to the base of the sulcus/pocket

SECONDARY OUTCOMES:
Bleeding on probing | Baseline and 3 months after treatment
  Sign of bleeding after gentle probing of the sulcus/periodontal pocket
Clinical attachment level | Baseline and 3 months after treatment
  The distance from the CEJ to the base of the sulcus/pocket
Oral Health Impact Profile-14 | Baseline and 3 months after treatment
  A questionnaire designed to determine oral health related quality of life consists of seven domains reflecting Functional limitation, Physical pain, Psychological discomfort, Physical disability, Psychological disability, Social disability, Handicap. Each domain composed of two questions and the scores calculation are based on a Likert scale (Never, Hardly ever, Occasionally, Often, Very often) which receive scores from 0 to 4. The higher total scores indicate worse oral health related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry/ University of Baghdad, Baghdad, Iraq